CLINICAL TRIAL: NCT04640389
Title: Rural-urban Disparities in the Nutritional Status of Younger Adolescents in Tanzania.
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: UNICEF (Other); Harvard University (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Lorraine Cordeiro, Associate Professor, University of Massachusetts, Amherst
Other Study IDs: 15-008
Record Dates: First submitted 2020-11-11; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Undernutrition; Stunting; Adolescent Development
MeSH Terms: conditions — Malnutrition; Growth Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urban: Urban adolescents living in Moshi District, Tanzania, who are between 10-14 years of age.
  Interventions: Other: Cross-sectional study/no intervention
- Rural: Rural adolescents living in Kilosa District, Tanzania, who are between 10-14 years of age.
  Interventions: Other: Cross-sectional study/no intervention

INTERVENTIONS:
Other: Cross-sectional study/no intervention — Cross-sectional study/no intervention.

SUMMARY:
Africa faces rapid urbanization, has the second highest population growth rate, makes up one-fifth of the world's youth population, and experiences stagnant rates of undernutrition. These challenges point to the need for country-specific data on rural-urban health disparities to inform development policies. This cross-sectional study examined disparities in body mass index-for-age-and-sex (BAZ) and height-for-age-and-sex z-scores (HAZ) among 1125 adolescents in Tanzania. Rural-urban disparities in nutritional status were significant and gendered. Findings confirm place of residence as a key determinant of BAZ, HAZ, and stunting among adolescents in Tanzania. Targeted gender-sensitive interventions among adolescents, particularly in rural areas, are needed to limit growth faltering and improve health outcomes.

DETAILED DESCRIPTION:
Africa faces rapid urbanization, has the second highest population growth rate, makes up one-fifth of the world's youth population, and experiences stagnant rates of undernutrition. These challenges point to the need for country-specific data on rural-urban health disparities to inform development policies. This cross-sectional study examined disparities in body mass index-for-age-and-sex (BAZ) and height-for-age-and-sex z-scores (HAZ) among 1125 adolescents in Tanzania. Pearson's chi-square tested associations between rural/urban residence and undernutrition (BAZ <-2SD), stunting (HAZ <-2SD), anthropometric, socioeconomic, and health indicators. Multivariate linear regression identified predictors of BAZ and HAZ.

Funding: UNICEF/ Tanzania; United States National Institute of Mental Health (R01 MH66801).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 10 and 14 years of age

Exclusion Criteria:

* Adolescents living away from the districts and not physically present at the time of the study

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This cross-sectional study merged and analyzed two independent samples of adolescents living in Tanzania. One study was conducted in Tanzania by Cordeiro et al. (2012) and the other was conducted in an urban setting by Carlson, Brennan, and Earls (2012); both conducted in 2004. The Kilosa/rural dataset was derived from a two-stage sampling plan for selection of villages and adolescents. The Moshi/urban dataset was derived from a two-stage sampling plan for a cluster randomized control trial (CRCT). From a total combined sample of 1476 adolescents aged 10-19 years across both datasets, 1237 met the age criterion for younger adolescents (10-14 years). The analytical sample for this study was 1125.
Sampling Method: Probability Sample
Enrollment: 1125 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index for age and gender z-scores | Two measures collected consequentially during a 30 minute time frame on the date of survey administration.
  Weight (Kg)/Height (M) squared compared to the WHO growth reference standard
Height for age and gender z-scores | Two measures collected consequentially during a 30 minute time frame on the date of survey administration.
  Height in meters for age and gender compared to the WHO growth reference standard
Undernutrition | Height and weight measures collected twice consequentially during a 30 minute time frame on the date of survey administration.
  Body Mass Index for age and gender z-scores < -2SD of the WHO growth reference standard
Stunting | Two measures of height in meters collected consequentially during a 30 minute time frame on the date of survey administration.
  Height (M) for age and gender z-scores < -2SD of the WHO growth reference

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Cordeiro, Ph.D., Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordeiro LS, Wilde PE, Semu H, Levinson FJ. Household food security is inversely associated with undernutrition among adolescents from Kilosa, Tanzania. J Nutr. 2012 Sep;142(9):1741-7. doi: 10.3945/jn.111.155994. Epub 2012 Jul 18. PMID 22810984
- [Background] Carlson M, Brennan RT, Earls F. Enhancing adolescent self-efficacy and collective efficacy through public engagement around HIV/AIDS competence: a multilevel, cluster randomized-controlled trial. Soc Sci Med. 2012 Sep;75(6):1078-87. doi: 10.1016/j.socscimed.2012.04.035. Epub 2012 May 24. PMID 22703885